CLINICAL TRIAL: NCT00582946
Title: Wide-Bandwidth Open Canal Hearing Aid For Better Multitalker Speech Understanding
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EarLens Corporation (Industry)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Suzy Levy, Ph.D., Director of Clinical, For Sunil Puria, Chief Scientist (no longer with company), EarLens Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: R43DC008499-01 (NIH); R44DC008499 (NIH)
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Results first posted 2016-10-03 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-09

CONDITIONS: Hearing Impairment
Keywords: Hearing Loss, Eardrum, Transducer, Hearing in Noise
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Magnetic Contact Hearing Aid (Experimental): Subjects were treated with a hearing aid which provided amplification intended to treat mild to moderate sensorineural hearing loss. Acute performance and safety assessed at 4 months compared to unaided baseline pre-treatment, followed by longer-term assessment of safety up to 10 months.
  Interventions: Device: Hearing Aid

INTERVENTIONS:
Device: Hearing Aid — Subjects were treated with a hearing aid which provided amplification intended to treat mild to moderate sensorineural hearing loss.

SUMMARY:
Our goal is to design and build a new hearing aid system, which mitigates the most common complaints that hearing aid users have. These include hearing in multi-talker situations, poor sound quality, unwanted whistling resulting from feedback, and a dislike of the sound of their own voice. Current efforts, with limited success, use signal processing methods rather than restoring more closely the normal auditory function. We plan to achieve our goal by reducing to practice three key enabling concepts. The first is to replace the current acoustic transducer with a non-acoustic mechanical output transducer that directly actuates the tympanic membrane (TM). This transducer, called the EarLens, floats on the tympanic membrane in a manner similar to the way a contract lens floats on the eye. The second is to increase the output bandwidth of the hearing aid. The third key concept is to place a wide-bandwidth microphone in the ear canal to capture the pinna diffraction cues similarly to the way the normal ear functions. Our central hypothesis is that a hearing aid that delivers amplified wide-bandwidth mechanical stimuli, directionally dependent cues, in an open canal configuration will perform better than conventional hearing aids when there are competing talkers in the background. First phase includes verification the capability of the system to deliver sufficient maximum equivalent pressure output (MEPO) to treat the degree of hearing loss in the target fitting range.

ELIGIBILITY:
Inclusion Criteria:

* Hearing loss less than 60 dB at any frequency, no conductive hearing loss

Exclusion Criteria:

* Collapsed ear canal, damaged or repaired middle ear, too much sensory hearing loss

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Puria, Principal Investigator — Ear Lens Corporation
Locations (1):
- Ear Lens Corporation, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No
Please see publication for summary results.

REFERENCES:
- [Result] Perkins R, Fay JP, Rucker P, Rosen M, Olson L, Puria S. The EarLens system: new sound transduction methods. Hear Res. 2010 May;263(1-2):104-13. doi: 10.1016/j.heares.2010.01.012. Epub 2010 Jan 29. PMID 20116419
- See also: Electromagnetic EarLens system published in Hearing Research — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2974567/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Magnetic Contact Hearing Aid
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Magnetic Contact Hearing Aid
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Maximum Effective Sound Pressure Level (MEPO)
Description: A primary outcome measure of interest is an estimate of the insitu maximum equivalent pressure output (MEPO) of the EarLens system, which represents the sound pressure level that would have to be applied at the eardrum (or tympanic membrane) to produce the same degree of tympanic membrane (TM) vibration that the EarLens system produces with the coil current set to its maximum value, and given the anatomical constraints on the coupling between the coil and magnet for a given subject. The target fitting range included hearing loss up to 60 decibels (dB) Hearing Level (HL). In order for the device to be an effective hearing aid for this target population, the maximum output of the device needs to be able to provide output and gain to treat this maximum hearing loss.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: decibels (dB) Sound Pressure Level (SPL)
Groups:
- Maximum Equivalent Pressure Output: Provision of amplification to treat sensorineural hearing loss with direct-drive hearing aid for acute evaluation of efficacy.
Arm/Group | Maximum Equivalent Pressure Output
Number analyzed (Participants) | 16
decibels (dB) Sound Pressure Level (SPL) | 95 (7)

ADVERSE EVENTS:
Time Frame: From treatment to study completion, up to 10 months.
Arm/Group | Magnetic Contact Hearing Aid
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes